CLINICAL TRIAL: NCT00952406
Title: A Multi Center Study to Validate a Condition-specific Measure of Sexual Health in Women With Pelvic Floor Disorders
Status: Completed | Type: Observational
Sponsor: International Urogynecological Society (Other)
Responsible Party: Principal Investigator, Rebecca G Rogers, Principal Investigator, International Urogynecological Society
Other Study IDs: IUGA -1 - 09
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Pelvic Floor Disorders; Sexual Dysfunction; Incontinence; Pelvic Organ Prolapse
Keywords: Pelvic Floor Disorders; Sexual Function; Incontinence; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Floor Disorders; Sexual Dysfunction, Physiological; Pelvic Organ Prolapse | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No Biospecimens are to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey of Women PFDs: Women with PFDs
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — This is a study to develop a survey for sexual health in women with pelvic floor dysfunction

SUMMARY:
Study Aims:

1. To validate a new measure of sexual function and activity in women with PFDs;
2. To establish the responsiveness to change of the new measure.

The investigators hypothesis is that the investigators can create a new questionnaire that accurately measures sexual health in women with pelvic floor disorders that improves on the already published questionnaires.

DETAILED DESCRIPTION:
600 women presenting for care to urogynecology clinics in the United States and England will be recruited to participate. They will give data regarding their physical exam, including measurements by the Pelvic Organ Prolapse Quantification exam and medical and surgical history. In addition, they will complete validated questionnaires including the Incontinence Severity Index, the Pelvic Floor Distress Inventory (short form) and question # 35 from the Epidemiology of Prolapse and Incontinence Questionnaire. All women will also complete two sexual health questionnaires; the Female Sexual Function Index and the Pelvic Organ Prolapse Urinary Incontinence Sexual Questionnaire (Revised). Women will receive standard care for their pelvic floor disorders. They will then be recontacted to repeat the same set of questionnaires to determine the responsiveness of the new measure. Reliability of the questionnaire will be measured by having a subset of women complete the questionnaire twice; a factor analysis will be performed to determine the underlying factor structure. Responses to the other QOL measures will be compared to those to the new instrument to establish validity.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients include age over 18 years.
* Not pregnant.
* Able to read/write and understand English.
* And, because this is a project to validate a measure of female sexual function, all subjects will be women.
* All women will be seeking care for PFD including urinary and anal incontinence and POP. Since data collection will primarily be by mail
* Women must have a stable and current address.

Exclusion Criteria:

* Women under the age of 18.
* Are pregnant or who are unable to read/write or understand English will not be eligible for participation.
* In addition, women with a diagnosis of vulvodynia, painful bladder syndrome, or chronic pelvic pain (defined as pelvic pain for greater than 6 months) as determined by the consenting physician will be excluded.
* Since this is a study to evaluate both sexual activity status as well as sexual function, women need not be sexually active to participate.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Goal to enroll approximately 800 women so that 600 surveys are available for evaluation of the sexual health of women with pelvic floor disorders presenting for urogynecological care in the United States or England
Sampling Method: Non-Probability Sample
Enrollment: 877 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study is the creation of a valid and reliable new measure of sexual health in women with pelvic floor disorders. | 3-5 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Rogers, MD, Principal Investigator — University of New Mexico Health Sciences Center
Locations (14):
- United States (9):
  - UCSD women's Pelvic Medicine Center, San Diego, California
  - Northwestern University Feinburg School of Medicine, Evanston, Illinois
  - MetroUrology, Minneapolis, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Women's Pelvic Speciality Care PC, Albuquerque, New Mexico
  - Center for Female Sexual Health, Cincinnati, Ohio
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - Genesis Health System, Zanesville, Ohio
  - Geisinger Health Systems, Danville, Pennsylvania
- United Kingdom (5):
  - Chelsea and Westminster Hospital, London
  - The Warrell Unit, Whitworth Park, Manchester
  - Northwick Park and St Marks Hospital, Middlesex
  - Royal Hallamshire Hospital, Sheffield
  - Mayday University Hospital, Surrey

REFERENCES:
- [Background] Rogers RG, Espuna Pons ME. The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR). Int Urogynecol J. 2013 Jul;24(7):1063-4. doi: 10.1007/s00192-012-1952-3. Epub 2013 Apr 30. No abstract available. PMID 23632797
- [Result] Kanter G, Jeppson PC, McGuire BL, Rogers RG. Perineorrhaphy: commonly performed yet poorly understood. A survey of surgeons. Int Urogynecol J. 2015 Dec;26(12):1797-801. doi: 10.1007/s00192-015-2762-1. Epub 2015 Jul 4. PMID 26142348
- [Result] Rockwood TH, Constantine ML, Adegoke O, Rogers RG, McDermott E, Davila GW, Domoney C, Jha S, Kammerer-Doak D, Lukacz ES, Parekh M, Pauls R, Pitkin J, Reid F, Ridgeway B, Thakar R, Sand PK, Sutherland SE, Espuna-Pons M. The PISQ-IR: considerations in scale scoring and development. Int Urogynecol J. 2013 Jul;24(7):1105-22. doi: 10.1007/s00192-012-2037-z. Epub 2013 Apr 30. PMID 23632799
- [Result] Rogers RG, Rockwood TH, Constantine ML, Thakar R, Kammerer-Doak DN, Pauls RN, Parekh M, Ridgeway B, Jha S, Pitkin J, Reid F, Sutherland SE, Lukacz ES, Domoney C, Sand P, Davila GW, Espuna Pons ME. A new measure of sexual function in women with pelvic floor disorders (PFD): the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR). Int Urogynecol J. 2013 Jul;24(7):1091-103. doi: 10.1007/s00192-012-2020-8. Epub 2013 Apr 30. PMID 23632798
- [Result] Pauls RN, Rogers RG, Parekh M, Pitkin J, Kammerer-Doak D, Sand P. Sexual function in women with anal incontinence using a new instrument: the PISQ-IR. Int Urogynecol J. 2015 May;26(5):657-63. doi: 10.1007/s00192-014-2563-y. Epub 2014 Nov 13. PMID 25392184